CLINICAL TRIAL: NCT07115563
Title: Effects of Targeted Amino Acid Supplementation for People With Parkinson's Disease on Amino Acid Profiles and Health Related Markers
Brief Title: Daily Amino Acid Supplementation for People With Parkinson's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cristina Colon-Semenza (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Cristina Colon-Semenza, Assistant Professor, University of Connecticut
Organization: University of Connecticut (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 25-02-219-910; B2025-0194 (Other Grant/Funding Number: USDA-NIFA)
Record Dates: First submitted 2025-07-29; First posted 2025-08-11 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Parkinson Disease (PD)
Keywords: Nutrition; Parkinson's disease; Amino acid supplements
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): The inert amino acid (alanine) will serve as an isonitrogenous control.
  Interventions: Dietary Supplement: Control (placebo)
- Targeted Amino Acid Supplement (Experimental): Blend of the essential amino acids (Leucine & Tryptophan), a conditionally essential amino acids (Arginine & Taurine), and non-essential amino acids (Glutamate & Tyrosine) designed to meet the unique nutritional needs of people with Parkinson's disease (PD).
  Interventions: Dietary Supplement: Targeted Amino Acid Supplement

INTERVENTIONS:
Dietary Supplement: Targeted Amino Acid Supplement — Blend of the essential amino acids (Leucine & Tryptophan), a conditionally essential amino acids (Arginine & Taurine), and non-essential amino acids (Glutamate & Tyrosine) designed to meet the unique nutritional needs of people with Parkinson's disease (PD).
  Arms: Targeted Amino Acid Supplement
Dietary Supplement: Control (placebo) — The inert amino acid (alanine) will serve as an isonitrogenous control.
  Arms: Control

SUMMARY:
The goal of this clinical trial is to learn if a tailored amino acid supplement works to help adults living with Parkinson's disease to improve nutrition, metabolic function, body composition, and physical and mental function. The main questions it aims to answer are:

Does the tailored amino acid supplement increase essential amino acids (nutritional status)?

Does the tailored amino acid supplement increase an antioxidant (complex amino acid) and decrease an amino acid associated with oxidative stress?

Does the tailored amino acid supplement improve physical and mental health compared to a placebo supplement?

Researchers will compare the tailored amino acid supplement to a placebo (a look-alike substance that contains no active ingredients) to see if the tailored amino acid supplements work to support health for people with Parkinson's disease.

Participants will:

Take the tailored amino acid supplement or a placebo every day for 6 months, visit the lab at baseline, after 3 months, and after 6 months for fasting blood draws, body composition assessment, and physical and mental health testing and keep a diary of their food intake and supplement intake.

DETAILED DESCRIPTION:
The purpose of this trial is to determine the effects of a targeted amino acid supplement (T-AA) specifically designed to correct characteristic amino acid deficiencies and meet the unique nutritional needs of people with Parkinson's disease (PD) on 1) plasma amino acid (AA) bioavailability, 2) metabolic function, 3) body composition, 4) physical function and 5) self-reported outcomes.

ELIGIBILITY:
Inclusionary Criteria:

* Male and Females.
* 60-80 Years.
* Previous diagnosis of idiopathic Parkinson's Disease by patient report.
* Use of dopamine replacement medication (e.g. levodopa) for at least 2 years.
* On a stable dose of dopamine replacement medication for at least 3 months with no plans for change in the next two months.

Exclusionary criteria

* Apparent cognitive impairment as determined by phone screening (Telephone Interview for Cognitive Status <29).
* Diagnosis of Parkinsonism or atypical Parkinson's Disease.
* Prescription of Dopamine antagonist.
* Any unstable medical condition.
* Any known bleeding disorder or current consumption of blood thinners.
* Use of Deep Brain Stimulation.
* Gastric or Bowel resection surgery.
* Contraindications to blood draw.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-31 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Amino Acid bioavailability (Lysine, Tryptophan, Arginine, Glutamate, Leucine, Taurine, Glutathione) | Baseline, 3 months, and 6 months
  Circulating amino acid concentrations will be measured from blood samples using high performance liquid chromatography using a solid phase column specifically designed to test amino acids (e.g. 00F-4435-E0, Phenomenex, USA) along with appropriate column guards (e.g. AJ0-7597 & KJ0-4282, Phenomenex, USA) and liquid phases. This analysis will be performed at the Laboratory of Mass Spectroscopy and Omics Analysis.
Oxidative stress | Baseline, 3 months, 6 months
  Oxidative stress will be measured using a total antioxidant power test (e.g. ab65329, ABCAM, USA). It is a quantitative bioassay and will be performed using the laboratory facilities.
Oxidative stress | Baseline, 3 months, and 6 months
  Oxidative stress will be assessed with reduced/oxidized glutathione assays (e.g. ab138881, ABCAM, USA). It is a quantitative bioassay and will be assessed using laboratory facilities.

SECONDARY OUTCOMES:
Body composition: Bioelectrical impedance | Baseline, 3 months, 6 months
  Body composition will be assessed using a multi-spectral bioelectrical impedance (Mediana i55, Mediana, South Korea). During this test participants will clean their feet and hands using a sanitary wipe and then stand barefoot on the impedance machine while holding two electrodes. Then a small and imperceivable multi-spectral electrical current will be sent between limbs which the machine will use to estimate the fat content and distribution based on the resistance (i.e., impedance) of this current.
Body composition: Ultrasound & Shear Wave Elastography (Tissue Organization & Fibrosis) | Baseline, 3 months, 6 months
  A trained (>20 hr. logged research scanning) ultrasound researcher will use an ultrasound (ACUSON Sequoia, Siemens Healthineers, USA) to assess muscle thickness of the primary knee extensors (quadriceps femoris) and the plantar flexors (gastrocnemius and soleus) as well as their tendons. Longitudinal panoramic 2D ultrasound will be used to measure muscle fascicle length and angle of each muscle. To assess tissue composition of these muscles shear-wave elastography will be used to measure localized muscle stiffness based on propagation of a concentrated acoustic shear (push-pull) wave applied to the center of the muscle.
Physical function: Physical activity | 7 days prior to baseline visit and 7 days after the 6-month visit
  Participants will be sent a research-grade activity monitor, Actigraph GT9X device, in the standard mail at their residence. After receiving the device, participants will engage in a telephone or virtual meeting with a research assistant to learn how to use the device. (approximately 30-40 minutes). Participants will be asked to wear the activity monitor for 7 days prior to the first baseline visit. They will be asked to continuously wear the device on their wrist for the 7 days. Participants will return the device in a pre-paid envelope. The same procedure will occur at the conclusion of the intervention for a post-intervention assessment.
Physical function: Balance (Mini Balance Evaluation System Test) | baseline, 3 months, 6 months
  This test assesses balance impairments across 14 items consisting of dynamic balance, anticipatory postural adjustments, reactive postural control, sensory orientation and dynamic gait. The total score ranges from 0 to 28, with each item scored on a scale from 0 to 2 with higher scores indicating better balance.
Physical function: Gait speed (4-meter walking test) | baseline, 3 months, 6 months
  This physical test measures the speed at which a person can walk for 4 meters which is related to overall functional ability. The patient is asked to walk at normal speed for 4 meters, while the evaluator records the time required for it. The gait speed is calculated dividing the distance (4m) by the time completed by the participant. The fastest of 2 trials is then recorded.
Physical function: Gait speed (10-meter walk test) | baseline, 3 months, 6 months
  This test measures the speed at which a person can walk for 10 meters. The participant will walk for 10 meters, divided by 2 initial meters of acceleration and 2 final meters for deacceleration. The walking speed during the central 6 meters is then recorded.
Physical function: Functional lower extremity strength (5 Times Sit to Stand Test) | baseline, 3 months, 6 months
  The Five Times Sit to Stand Test is a physical test for measuring functional strength in the lower limbs. For this test, the participant must stand up and sit down on an armless chair with their arms crossed on their chest as fast as possible 5 times. A practice trial is permitted before the test trial.
Physical function: Grip strength | baseline, 3 months, 6 months
  Bilateral grip strength will be assessed with the use of a handheld dynamometer. For this test the participant must be seated on a chair, with the assessed limb at 90º of elbow flexion and holding the dynamometer in a neutral wrist position. Two sub-maximal trials at 50% and 70% of the Maximal voluntary Isometric grip contraction will be performed as a warmup. Then, 3 maximal trials separated by 1 minute of rest will be performed. If there is a 5% or bigger difference in strength for any trial, a fourth attempt must be completed. The highest value obtained for each limb is recorded.
Physical function: Maximal voluntary isometric contraction | baseline, 3 months, 6 months
  In these tests participants will be seated in an isometric dynamometer (Biodex System 4, Biodex, USA) with their body and dynamometers positioned according to manufacturer instructions. In these positions participants will perform three submaximal practice isometric contractions (~25%, 50%, and 75% maximal effort) and then 5 maximal effect isometric contractions with each contraction separated 1 min of rest.
Self-reported outcome: Quality of Life (Parkinson Disease Questionnaire-39) | baseline, 3 months, 6 months
  This questionnaire assesses the difficulties that people with PD experience across 8 dimensions of daily living; Activities of Daily Living, Attention & Working Memory, Cognition, Communication, Depression, Functional Mobility, Quality of Life, Social Relationships and Social Support. The score ranges from 0-100 with higher scores indicating worse quality of life.
Self-reported outcome: Fatigue (Parkinson's Fatigue Scale) | baseline, 3 months, 6 months
  This is a 16-Item patient-rated questionnaire that quantifies fatigue in people with PD. The scores range from 16 to 80 with higher scores indicating higher levels of fatigue.
Self-reported outcome: Sleep (Scales for Outcomes in Parkinson disease- Sleep, nighttime sleep) | baseline, 3 months, 6 months
  This is a patient-reported questionnaire that assess nighttime sleep across 5 items in patients with Parkinson's disease. The score ranges from 0-15 with higher scores indicating worse sleep.
Self-reported outcome: Sleep (Scales for Outcomes in Parkinson disease- Sleep, daytime sleepiness) | Baseline, 3 months, 6 months
  This is a patient-reported questionnaire that assess daytime sleepiness across 6 items in patients with Parkinson's disease. The score ranges from 0-18 with higher scores indicating more daytime sleepiness.
Self-reported outcome: Sleep (Scales for Outcomes in PD-Sleep, Global sleep quality) | Baseline, 3 months, 6 months
  This is a patient-reported questionnaire that assess the individual's global assessment of nighttime sleep with one item in patients with Parkinson disease. The score ranges from 0-6 with higher scores indicating worse global sleep quality.
Self-reported outcome: Mood (Profile of Mood State) | baseline, 3 months, 6 months
  This an assessment of current mood state. It is a 40-item self-report survey that evaluates the degree to which a participant is feeling a selected emotion at the moment. The score ranges from -30 to 200 with higher scores indicating worse mood.
Self-reported outcome: Anxiety (Beck Anxiety Inventory) | baseline, 3 months, 6 months
  This is an assessment of somatic and cognitive symptoms of anxiety. It consists of 21 items in the form of self-reported questionnaire. The score ranges from 0-63 with higher scores indicating higher levels of anxiety.
Self-reported outcome: Motivation (Behavioral Regulation in Exercise Questionnaire-2) | baseline, 3 months, 6 months
  This is the most used measure of motivators for exercise. It is a 19-item survey that evaluates the stages of motivation to exercise. This includes amotivation, external regulation, introjected regulation, identified regulation, and intrinsic regulation. The score ranges from -24 to +20 with higher scores indicating increased motivation.
Self-reported outcome: Depression (Geriatric Depression Scale-short form) | baseline, 3 months, 6 months
  This is a 15-item self-report measure of depression in older adults. Scores range from 0-15 with higher scores indicating more severe depression.
Insulin sensitivity | baseline, 3 months, 6 months
  Blood drawn will be used to analyze blood glucose. A test strip will be inserted into a glucose meter and a small sample of blood will be applied. The blood glucose level will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Connecticut, Storrs, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD used in the results publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Beginning 1 year after publication and ending 3 years after the publication of results
Access Criteria: A proposal for planned analyses must be submitted, a data sharing agreement must be signed, and documents must be submitted to the PIs, Dr. Earp and Dr. Colón-Semenza via email. Requests will be reviewed by the PIs to determine eligibility. Eligible individuals must have expertise in Parkinson disease, nutrition, and/or oxidative stress and antioxidant capacity, and have a position at a research institution with a dissemination plan of making their results publicly available through peer-reviewed publications. This data will not be shared with commercial entities.

REFERENCES:
- [Background] Earp JE, Colon-Semenza C, LoBuono DL. Considerations for developing a targeted amino acid supplement for people with Parkinson's disease that promotes health while accounting for pathophysiology and medication interference. Nutr Rev. 2023 Jul 10;81(8):1063-1076. doi: 10.1093/nutrit/nuad008. PMID 36809398